CLINICAL TRIAL: NCT00916175
Title: Randomized Double Blind Factorial Assay, Aloe Vera (AV) And/Or Cnidoscolus Chayamansa (CC) Versus Placebo, Reduction Of High Blood Glucose In Women With Metabolic Syndrome
Brief Title: Metabolic Syndrome and Functional Food
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Lilia Csrdenas-Ibarra, MD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EN_LC_P134
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2009-07

CONDITIONS: Metabolic Syndrome
Keywords: hyperglycemia; overweight; functional food; aloe vera; cnidoscolus chayamansa
MeSH Terms: conditions — Metabolic Syndrome; Hyperglycemia; Overweight | interventions — Aloe vera gel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- P1&P2 (Placebo Comparator): Food product P1&P2 is composed of: placebo1(mimic aloe vera gel) 30ml and placebo2 (mimic Cnidoscolus chayamansa infusion) 200ml;
  Interventions: Dietary Supplement: P1&P2
- P1&CC (Experimental): Food Product P1&CC contains: placebo1 (mimics liquified aloe vera gel) 30ml and Cnidoscolus Chayamansa infusion 200ml;
  Interventions: Dietary Supplement: P1&CC
- AG&P2 (Experimental): Food product AG&P2 contains (liquified aloe vera gel) 30ml and placebo2 (mimic CC infusion) 200ml.
  Interventions: Dietary Supplement: AG&P2
- AG&CC (Experimental): Food product AG&CC is composed of: liquified aloe vera gel 30ml and Cnidoscolus Chayamansa infusion 200ml
  Interventions: Dietary Supplement: AG&CC
- TA (concentrated 5:1 aloe vera gel) (Experimental): Food product TA contains concentrated 5:1 aloe vera gel by total process30 ml and purified water 200 ml.
  Interventions: Dietary Supplement: TA (concentrated 5:1 aloe vera gel)
- P3 (Placebo Comparator): Food product Placebo 3 contains stabilizers and preservative used for TA 30 ml and purified water 200 ml.
  Interventions: Dietary Supplement: P3

INTERVENTIONS:
Dietary Supplement: P1&P2 — * First period (4 weeks) intake food product P1&P2 (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet
  * Second period, cross over from AG&CC group, 4 weeks intake food product P1&P2 (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet
  Other Names: Placebo 1 and Placebo 2
  Arms: P1&P2
Dietary Supplement: P1&CC — * First period (4 weeks) intake food product P1&CC (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet.
  * Second period, cross over from AG&P2 group, 4 weeks intake food product P1&CC (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet.
  Other Names: Placebo 1 and Cnidoscolus Chayamansa infusion
  Arms: P1&CC
Dietary Supplement: AG&P2 — * First period (4 weeks) intake food product AG&P2 (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet.
  * Second period, cross over from P1&CC group, 4 weeks intake food product AG&P2 (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet
  Other Names: Aloe Vera Gel and Placebo 2
  Arms: AG&P2
Dietary Supplement: AG&CC — * First period (4 weeks) intake food product AG&CC (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet
  * Second period, cross over from P1&P2 group, 4 weeks intake food product AG&CC (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet
  Other Names: Aloe Vera gel and Cnidoscolus Chayamansa infusion; Sabila & Chaya infusion
  Arms: AG&CC
Dietary Supplement: TA (concentrated 5:1 aloe vera gel) — * First period (4 weeks) intake food product TA (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet.
  * Second period, cross over from P3 group, 4 weeks intake food product TA (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet.
  Other Names: Total Aloe concentrated 5:1 aloe vera gel by total process
  Arms: TA (concentrated 5:1 aloe vera gel)
Dietary Supplement: P3 — * First period (4 weeks) intake food product P3 (in lemon gelatin 230 ml before breakfast) plus 1500 kilo calories diet.
  * Second period, cross over from TA group, 4 weeks intake food product P3 (in lemon gelatin 230 ml before breakfast and 230 ml after supper) plus 1500 kilo calories diet.
  Other Names: Placebo 3
  Arms: P3

SUMMARY:
High blood sugar and adiposity are part of Metabolic syndrome (about 24% of adults harbor it). The main approach, weight reduction, is often unattainable. Aloe Vera (barbadensis) (AV) and cnidoscolus chayamansa (McVaugh)(CC) are two vegetables that seem to have an effect on blood glucose and body weight.

The study aims to determine if the intake of aloe gel and/or Chaya infusion can reduce high blood sugar in adult women with pre-diabetes (Metabolic Syndrome).

Methods: A Factorial assay, double blind, cross-over-controlled with random assignment, to four treatments: AV and CC, AV and Placebo 1, Placebo 2 and CC, and Placebo 1 and Placebo 2, at the outpatient clinic of the university Hospital and a community clinic.

Two treatment periods of 4 weeks intermediated by one week for wash-out.

ELIGIBILITY:
Inclusion criteria:

* Adult women living in Monterrey, Mexico with at least three of the following:

  * waist line equal or larger than 88 cm
  * fasting blood sugar between 100-140 mg/dL without symptoms or known glucose intolerance or diabetes treated only with diet
  * known high blood pressure or 2/3 readings systolic > 130 mmHg, diastolic > 85
  * HLD < 50 mg/dL or triglycerides > 150 mg/dL

Exclusion Criteria:

* Pregnancy or nursing
* On anti-diabetic agents
* Diabetic symptoms or advanced DM complications
* Severe behavioral problems

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Reduction of elevated blood sugar (HbA1c) by Immunoturbidimetric test (One-HbA1c FS) via Star-Dust MC15; both from Diagnostic systems international (DiaSys); its coefficient of variation was 1.6%. | baseline, and at the end of each of 2 treatment periods of 4 weeks

SECONDARY OUTCOMES:
Significant changes on hematic biometry and liver function test and evaluation of any symptoms reported. | baseline, and after four weeks of treatment or sooner if needed
Tolerance assessed by weekly inquiry of effort needed to take the product, wellbeing, energy, gastrointestinal complains, control of appetite and general complaints. | after each week taking the product

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Cardenas-Ibarra, MD, Principal Investigator — Endocrinology, University Hospital, Universidad Autonoma de Nuevo Leon; Jesus Z Villarreal-Perez, MD, Study Chair — Endocrinology, University Hospital, Universidad Autonoma de Nuevo Leon
Locations (2):
- Mexico (2):
  - Fomerrey 19 Community Clinic, Guadalupe, Nuevo León
  - Endocrinology, Outpatient clinic of University Hospital UANL, Monterrey, Nuevo León